CLINICAL TRIAL: NCT07041723
Title: Online Assessment and Enhancement of Auditory Perception for Speech Sound Errors: BiOfeedback, Online for Sibilant Treatment
Brief Title: BiOfeedback, Online for Sibilant Treatment
Acronym: BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-21-2137-Study 5; 2R15DC019775-02 (NIH)
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Speech Sound Disorder
Keywords: speech intervention; biofeedback; articulation disorder; lisp
MeSH Terms: conditions — Speech Sound Disorder; Articulation Disorders

STUDY DESIGN:
Intervention Model Description: For all treatment sessions, the participant and SLP will meet in a secure videoconference room. Participants will be provided with a standard headset with microphone (Plantronics Blackwire C3225) to capture their voice as input to the SonaSpeech II software running the SonaMatch real time FFT function. Information about the distribution of energy across the frequency range from the FFT spectrum has been found to reliably differentiate /s/ from other fricatives; clinically, this can be translated to differentiated perceptually accurate /s/ from misarticulated productions. Participants will view a real-time FFT spectrum and will be cued to match a visual target for /s/ where the spectral energy is concentrated to the right side of the display, primarily in the 5000-10,000 Hz region of the spectrum. Other aspects of the treatment protocol will follow the current research team's published guidelines for biofeedback intervention, modified for /s/ targets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual acoustic biofeedback (Experimental): Visual-acoustic biofeedback using the the SonaSpeech II software running the Sona Match module with the real-time FFT function.
  Interventions: Behavioral: Visual-acoustic biofeedback for Sibilants

INTERVENTIONS:
Behavioral: Visual-acoustic biofeedback for Sibilants — Participants will view a real-time FFT spectrum and will be cued to match a visual target for /s/ where the spectral energy is concentrated to the right side of the display, primarily in the 5000-10,000 Hz region of the spectrum. Practice will occur in blocks of 10 consecutive trials on the same item (e.g., 10 /sa/), after which a new item will be addressed (e.g., 10 /se/). Within each block, the clinician will provide qualitative (knowledge of performance) feedback as prompted by the research team's custom open-source software, Challenge Point Program (CPP). The CPP software prompts clinician actions such as delivery of knowledge of performance (KP) feedback. Following each block of ten trials, the software automatically tallies the scores entered by the clinician and uses the summed scores to make adaptive changes in practice difficulty.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of sibilant biofeedback treatment delivered via telepractice in six children ages 8:0-17;11 who present with distortions of /s/. The main questions it aims to answer are:

* Primary hypothesis: Biofeedback treatment for sibilants delivered via telepractice will produce positive gains compared to a no-treatment baseline phase.
* Secondary hypothesis: Participants will experience positive changes in social-emotional well-being after receiving biofeedback treatment for sibilants as reported by the participants and their guardians.

Following the initial evaluation, participants will be randomly assigned to transition from baseline to treatment at one of seven possible points, ranging from 4-10 baseline sessions in which /s/ production will be probed but not treated. All participants will then receive 20, 1-hour biofeedback treatment sessions over 10 weeks with a certified Speech-Language Pathologist via teletherapy, followed by three maintenance sessions.

DETAILED DESCRIPTION:
Study 2 will evaluate children with residual speech sound disorder affecting /s/ (n = 6). Both male and female children will be recruited. Participants must be between 8;0 and 17;11 years of age at the time of enrollment.

Randomization. Following the initial evaluation to determine eligibility, participants will be randomly assigned to transition from the baseline to the treatment condition at one of 7 possible points, ranging from 4 to 10 baseline sessions in which /s/ production will be probed but not treated. All participants will then receive 20 sessions of /s/ production training over 10 weeks, followed by 3 maintenance sessions.

Intervention Delivery. All treatment will be provided on an individual basis by a certified speech-language pathologist. Treatment will be delivered over Zoom videoconference calls using a unique password-protected room for each participant. In the beginning of each session a standard probe eliciting /s/ in various contexts at the sentence, word and syllable levels will be elicited. Following the /s/ probes, the session will consist of relatively unstructured, highly interactive prepractice for 10 minutes, which is designed to provide instruction on the phonetic requirements for /s/ and shaping strategies to transform the child's current productions into accurate /s/. The remainder of the session will elicit up to 150 syllables/words or 40 minutes of practice, whichever occurs first. Practice will occur in blocks of 10 consecutive trials on the same item (e.g., 10 /sa/), after which a new item will be addressed (e.g., 10 /se/). Within each block, the clinician will provide qualitative (knowledge of performance) feedback as prompted by the research team's custom open-source software, Challenge Point Program (CPP). The CPP software prompts clinician actions such as delivery of knowledge of performance (KP) feedback, promoting increased fidelity in treatment implementation both within and across sites. It also enables systematic changes in practice difficulty based on participant performance, as follows: after the software presents a stimulus and the participant attempts to produce it, the clinician scores the response as 0 or 1 based on their clinical impression of an incorrect or correct production of /s/. Following each block of ten trials, the software automatically tallies the scores entered by the clinician and uses them to make adaptive changes in practice difficulty. When a participant demonstrates at least 80% cumulative accuracy at the session level, the participants will be advanced from syllable to word-level practice; if the cumulative session-level accuracy drops below 50%, the participants will be dropped back to the syllable level to decrease difficulty. In word-level practice, parameters are adjusted on a rotating basis so that as accuracy increases, either the frequency of feedback is reduced (80%-50%-20%-0%), clinician models are faded, or word shapes increase in complexity. Qualitative feedback (either biofeedback or verbal clinician feedback) will begin at 80% of trials and, contingent upon the participant's performance, will be systematically decreased to 0% .

ELIGIBILITY:
Inclusion Criteria:

* Age between 8;0 and 17;11 years at the time of enrollment
* English as the dominant language (must have begun learning English by age 3, per parent report)
* Passes pure-tone hearing screening at 30 dB hearing level
* Passes brief examination of oral structure and function
* Less than 30% accuracy, based on consensus across 2 trained listeners, on a probe list eliciting fricative /s, z/ in various phonetic contexts at the word level
* No more than 3 sounds other than /s/ in error on the Goldman-Fristoe Test of Articulation-3 (GFTA-3)
* Diagnosis of ADHD, learning disability, dyslexia, or neurodiversity is admissible if participant meets cutoff scores on evaluation day 1
* History of CAS is admissible if participant meets cutoff scores on evaluation day 1
* Braces and removable retainers are admissible
* Access to a laptop or desktop computer and a quiet space for study sessions

Exclusion Criteria:

* Scaled score of 7 or higher on the Recalling Sentences and Formulated Sentences subtests of the Clinical Evaluation of Language Fundamentals-5 (CELF-5)
* History of permanent hearing loss (temporary hearing loss due to otitis media, including recurrent OM/tubes, is admissible)
* History of developmental disorder (e.g., Down syndrome, cerebral palsy)
* History of major brain injury, surgery, or stroke in the past year (mild concussion is admissible)
* Active diagnosis of epilepsy or other neurological disorder (permissible if well-controlled for at least 6 months)
* Current diagnosis of voice or fluency disorder
* Current presence of orthodontia that crosses the palate (braces and removable retainers are admissible)
* Lack of access to a laptop or desktop computer and a quiet space for study sessions

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Perceptually rated accuracy of /s/ production | Standard word probes will be elicited at baseline and post treatment (after 20 weeks).
  To assess generalization of perceptual training to production, participants will be assessed with standard probes administered in the first three baseline sessions , at the start of each treatment session and in three post-treatment maintenance sessions. Probes will elicit 60 words [considered the primary target], containing /s, z/ in various phonetic contexts. Stimuli in each probe will be presented individually in randomized order. No auditory models will be provided; for children with reading difficulty, semantic cues will be provided to elicit the intended word. Individual words will be isolated from the audio record of each word probe and presented in randomized order for binary rating (correct/incorrect) by 4 trained listeners who are blind to treatment condition and time point (but will see the written representation of each target word). The proportion of "correct" ratings for each token will be used as the measure of perceptually rated accuracy.

SECONDARY OUTCOMES:
Survey evaluating impacts of treatment on participants' socio-emotional well-being | The survey will be administered at baseline and post-treatment (after 20 weeks).
  This 11-item survey, which asks parents to report the impact of speech disorder on the child's social, emotional, and academic well-being, was validated in a published study by members of the research team. An impact score, calculated as described in the research team's previous research, will be used as the primary measure of socio-emotional well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Montclair State University, Bloomfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hitchcock ER, Ochs LC, Swartz MT, Leece MC, Preston JL, McAllister T. Tutorial: Using Visual-Acoustic Biofeedback for Speech Sound Training. Am J Speech Lang Pathol. 2023 Jan 11;32(1):18-36. doi: 10.1044/2022_AJSLP-22-00142. Epub 2023 Jan 9. PMID 36623212
- [Background] Shriberg, L.D., R. Paul, and P. Flipsen, Childhood speech sound disorders: From crow to the postgenomic era. Speech sound disorders in children, 2009: p. 1-33.
- [Background] Kraljevic JK, Matic A, Dokoza KP. Telepractice as a Reaction to the COVID-19 Crisis: Insights from Croatian SLP Settings. Int J Telerehabil. 2020 Dec 8;12(2):93-104. doi: 10.5195/ijt.2020.6325. PMID 33520098
- [Background] Whitehead E, Dorfman V, Tremper G, Kramer A, Sigler A, Gosman A. Telemedicine as a means of effective speech evaluation for patients with cleft palate. Ann Plast Surg. 2012 Apr;68(4):415-7. doi: 10.1097/SAP.0b013e31823b6897. PMID 22421491
- [Background] Lincoln M, Hines M, Fairweather C, Ramsden R, Martinovich J. Multiple stakeholder perspectives on teletherapy delivery of speech pathology services in rural schools: a preliminary, qualitative investigation. Int J Telerehabil. 2015 Jan 29;6(2):65-74. doi: 10.5195/IJT.2014.6155. eCollection 2014 Fall. PMID 25945230
- [Background] Wales D, Skinner L, Hayman M. The Efficacy of Telehealth-Delivered Speech and Language Intervention for Primary School-Age Children: A Systematic Review. Int J Telerehabil. 2017 Jun 29;9(1):55-70. doi: 10.5195/ijt.2017.6219. eCollection 2017 Spring. PMID 28814995